CLINICAL TRIAL: NCT02134119
Title: Echinacea-based Supplement Does Not Improve Markers of Performance in Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Georgia (Other)
Responsible Party: Principal Investigator, Jamie Cooper, Assistant Professor, University of Georgia
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: BRL-23C403; BRL-23C403 (Other Grant/Funding Number: Biomedical Research Laboratories, (grant #23C403))
Record Dates: First submitted 2014-05-02; First posted 2014-05-08 (Estimated); Results first posted 2017-01-05 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2016-11

CONDITIONS: Ineffective Erythropoiesis
Keywords: dietary supplement; endurance athletes; VO2max; red blood cells
MeSH Terms: interventions — Sugars

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Echinacea-based dietary supplement (Experimental): Echinacea-based dietary supplement 8,000mg/day or 16,000mg/day by mouth for 35-days
  Interventions: Dietary Supplement: Echinacea-based dietary supplement
- Sugar pill (Placebo Comparator): Placebo given 8,000mg/day by mouth
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: Echinacea-based dietary supplement — Echinacea-based dietary supplement given at 8,000mg/day or 16,000 mg/day by mouth
  Arms: Echinacea-based dietary supplement
Drug: Placebo — Sugar pill manufactured to mimic dietary supplement
  Other Names: Sugar pill manufactured to mimic dietary supplement
  Arms: Sugar pill

SUMMARY:
The purpose of this study was three-fold. We wanted to (1) determine if supplementation with an echinacea-based dietary supplement (ECH) would increase several blood parameters that could affect oxygen carrying capacity in the body, (2) determine if ECH would increase VO2max in trained endurance athletes, and (3) examine the effectiveness of two different doses of the ECH on all outcome variables. We hypothesized that supplementation with ECH would increase oxygen carrying capacity (as measured by RBCs, EPO, ferritin, hemoglobin (Hb), and hematocrit (Hct) levels), improve VO2max, and that the maximum dose would be most effective at increasing these outcomes.

DETAILED DESCRIPTION:
The supplement industry is a multi-billion dollar industry with many of the products targeted toward athletes and achieving optimal performance. Historically, endurance athletes have used a number of methods to try to increase erythrocyte (red blood cell-RBC) production in attempts to boost oxygen carrying capacity and perform better during aerobic exercise. A number of growth factors in the body can stimulate RBC production including erythropoietin (EPO). EPO is the primary growth factor that promotes the formation and release of RBCs from bone marrow. Although EPO itself is a banned substance, supplement companies have sought other means by which they can increase EPO production in the body in order to stimulate RBC synthesis. One natural product toted to stimulate EPO production is Echinacea and can be found in the product EPO-Boost™. Our global hypothesis is that supplementation of EPO-Boost™ will be an effective way to increase oxygen carrying capacity and improve maximal oxygen consumption in adult endurance athletes.

We will test whether EPO-Boost™ affects EPO levels, a number of blood parameters, and VO2max (maximal aerobic capacity) by recruiting 40 trained endurance athletes (20 males and 20 females). To be included, subjects must already be performing aerobic exercise at least 4 days per week for a minimum of one hour each day. Participants will be randomly assigned (within gender) to either the placebo (n=20) or supplement group (n=20). A 25% dropout rate may be expected in both genders, therefore we are recruiting a subject number of 40 participants to ensure that at least 30 subjects will complete the study. All participants will be blinded as to whether they are receiving the placebo or the supplement. Participants will report to the Human Nutrition Lab (HNL) and the Exercise Physiology Lab for baseline testing. Height, body weight, body composition, and blood samples will be obtained. Participants will then answer questions regarding their current and usual exercise patterns. These questions will address the type, frequency, duration, and intensity of exercise. Finally, participants will perform a VO2max test in the Exercise Physiology Lab. After baseline testing the participants will be given a supply of either EPO-Boost™ or placebo along with extra capsules. The subjects will not know whether they are receiving the product or the placebo. Participants will also be asked to consume a multivitamin pill daily for the entire 35-day intervention period. Finally, participants will be asked to keep an exercise log during the 35-day intervention documenting type, duration, intensity, and days of exercise in order for research personnel to ensure that exercise training is not changing. The capsule and exercise logs will be collected at days 14 and 35.

Blood collected during all 3 visits will be analyzed for EPO, ferritin, RBCs, white blood cells, hemoglobin, hematocrit, mean corpuscular volume, mean corpuscular hemoglobin, and mean corpuscular hemoglobin concentration. We will assess changes in blood parameters and VO2max to determine whether 35 days of EPO-Boost™ supplementation improves blood parameters or maximal aerobic capacity compared to placebo controls.

ELIGIBILITY:
Inclusion Criteria:

* Male and female endurance athletes between the ages of 18-44
* Normal body mass index (BMI) between 18.5-24.9kg/m2.
* Individuals must currently be performing aerobic exercise at least 4 days per week for a minimum of 60 minutes at each session.
* They must also be willing to maintain their current training regimen through the course of the study.

Exclusion Criteria:

* Any changes in altitude during the study (where they are living or training)
* Recent altitude training or use of a hypobaric chamber (within the last 6 months)
* Any other supplements or ergogenic aids (excluding multivitamins)
* Any participant who will be changing their current exercise training program during the study (includes changes in volume, frequency, or intensity)
* If any participant is pregnant, breastfeeding, or planning to become pregnant before this study would finish
* Any blood transfusions or blood donation in the past 16 weeks
* Any chronic diseases such as cardiovascular disease, renal disease, or diabetes
* Any condition that affects their ability to perform maximal exercise

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2012-01; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jamie A Cooper, Ph.D., Principal Investigator — Texas Tech University
Locations (1):
- Texas Tech University - Department of Nutritional Sciences, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Whitehead MT, Martin TD, Scheett TP, Webster MJ. The effect of 4 wk of oral echinacea supplementation on serum erythropoietin and indices of erythropoietic status. Int J Sport Nutr Exerc Metab. 2007 Aug;17(4):378-90. doi: 10.1123/ijsnem.17.4.378. PMID 17962712

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Echinacea-based Dietary Supplement | Sugar Pill
Started | 30 | 15
Completed | 30 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Echinacea-based Dietary Supplement | Sugar Pill | Total
Number analyzed (Participants) | 30 | 15 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.6 (7.6) | 29.9 (7.7) | 27.0 (7.8)
Gender [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 22 | 8 | 30

OUTCOME MEASURES:

1. Primary Outcome: VO2 Max
Description: A maximal graded exercise test on a treadmill (TrackMaster, TMX 425, Newton, KS) was used to determine VO2max using the modified Balke protocol. During the treadmill test, expired O2 and CO2 were continually measured using an open circuit metabolic measurement system (MedGraphics Ultima, CardioO2, St. Paul, MN). Participants performed a 5-minute warm-up on a treadmill at 0% grade. After the warm-up, the treadmill speed was then increased until participants were at 75% of their age-predicted maximal heart rate. Once this steady-state HR was achieved, the speed was kept constant while the grade increased by 2.5% every two minutes until volitional exhaustion. Criteria for ensuring that participants achieved VO2max in this study were achieving at least two of the following objective criteria: obtaining at least 90% of age-predicted max HR, a respiratory exchange ratio above 1.05, and/or a plateau in the VO2 response to exercise.
Time Frame: 0-days (baseline)
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | Echinacea-based Dietary Supplement | Sugar Pill
Number analyzed (Participants) | 30 | 15
ml/kg/min | 55.1 (6.6) | 56.7 (6.7)

2. Primary Outcome: VO2 Max
Description: as for outcome 1
Time Frame: 35-days
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | Echinacea-based Dietary Supplement | Sugar Pill
Number analyzed (Participants) | 30 | 15
ml/kg/min | 55.6 (7.6) | 57.8 (8.3)

3. Secondary Outcome: Hematological Measures - Red Blood Cells
Description: as measured by red blood cells (RBCs) at day 0 (baseline), day 14 (mid-intervention) and day 35 (post-intervention)
Time Frame: 0 days (baseline)
Measure: Mean (Standard Deviation); unit: M/uL
Arm/Group | Echinacea-based Dietary Supplement | Sugar Pill
Number analyzed (Participants) | 30 | 15
M/uL | 4.6 (0.6) | 4.6 (0.4)

4. Secondary Outcome: Hematological Measures - Red Blood Cells
Description: as measured by red blood cells (RBCs) at day 0 (baseline), day 14 (mid-intervention) and day 35 (post-intervention)
Time Frame: 14 days (mid-intervention)
Measure: Mean (Standard Deviation); unit: M/uL
Arm/Group | Echinacea-based Dietary Supplement | Sugar Pill
Number analyzed (Participants) | 30 | 15
M/uL | 4.6 (0.5) | 4.6 (0.45)

5. Secondary Outcome: Hematological Measures - Red Blood Cells
Description: as measured by red blood cells (RBCs) at day 0 (baseline), day 14 (mid-intervention) and day 35 (post-intervention)
Time Frame: 35 days
Measure: Mean (Standard Deviation); unit: M/uL
Arm/Group | Echinacea-based Dietary Supplement | Sugar Pill
Number analyzed (Participants) | 30 | 15
M/uL | 4.92 (0.6) | 4.6 (0.4)

6. Secondary Outcome: Hematological Measures - Erythropoietin
Description: as measured by erythropoietin (EPO) at day 0 (baseline), day 14 (mid-intervention) and day 35 (post-intervention)
Time Frame: 0 days (baseline)
Measure: Mean (Standard Deviation); unit: mU/mL
Arm/Group | Echinacea-based Dietary Supplement | Sugar Pill
Number analyzed (Participants) | 30 | 15
mU/mL | 7.2 (2.7) | 9.7 (3.1)

7. Secondary Outcome: Hematological Measures - Erythropoietin
Description: as measured by erythropoietin (EPO) at day 0 (baseline), day 14 (mid-intervention) and day 35 (post-intervention)
Time Frame: 14 days (mid-intervention)
Measure: Mean (Standard Deviation); unit: mU/mL
Arm/Group | Echinacea-based Dietary Supplement | Sugar Pill
Number analyzed (Participants) | 30 | 15
mU/mL | 7.3 (2.9) | 9.6 (2.5)

8. Secondary Outcome: Hematological Measures - Erythropoietin
Description: as measured by erythropoietin (EPO) at day 0 (baseline), day 14 (mid-intervention) and day 35 (post-intervention)
Time Frame: 35 days
Measure: Mean (Standard Deviation); unit: mU/mL
Arm/Group | Echinacea-based Dietary Supplement | Sugar Pill
Number analyzed (Participants) | 30 | 15
mU/mL | 7.1 (2.9) | 9.8 (2.2)

9. Secondary Outcome: Hematological Measures - Ferritin
Description: as measured by ferritin at day 0 (baseline), day 14 (mid-intervention) and day 35 (post-intervention)
Time Frame: 0 days (baseline)
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Echinacea-based Dietary Supplement | Sugar Pill
Number analyzed (Participants) | 30 | 15
ng/mL | 52.4 (47.3) | 69.8 (70.7)

10. Secondary Outcome: Hematological Measures - Ferritin
Description: as measured by ferritin at day 0 (baseline), day 14 (mid-intervention) and day 35 (post-intervention)
Time Frame: 14 days (mid-intervention)
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Echinacea-based Dietary Supplement | Sugar Pill
Number analyzed (Participants) | 30 | 15
ng/mL | 50.6 (46.2) | 59.4 (52.0)

11. Secondary Outcome: Hematological Measures - Ferritin
Description: as measured by ferritin at day 0 (baseline), day 14 (mid-intervention) and day 35 (post-intervention)
Time Frame: 35 days
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Echinacea-based Dietary Supplement | Sugar Pill
Number analyzed (Participants) | 30 | 15
ng/mL | 54.0 (41.0) | 51.7 (45.7)

12. Secondary Outcome: Hematological Measures - Hematocrit
Description: as measured by hematocrit (Hct) at day 0 (baseline), day 14 (mid-intervention) and day 35 (post-intervention)
Time Frame: 0 days (baseline)
Measure: Mean (Standard Deviation); unit: percent of red blood cells in blood
Arm/Group | Echinacea-based Dietary Supplement | Sugar Pill
Number analyzed (Participants) | 30 | 15
percent of red blood cells in blood | 41.7 (3.4) | 43.1 (3.5)

13. Secondary Outcome: Hematological Measures -Hematocrit
Description: as measured by hematocrit (Hct) at day 0 (baseline), day 14 (mid-intervention) and day 35 (post-intervention)
Time Frame: 14 days (mid-intervention)
Measure: Mean (Standard Deviation); unit: percent of red blood cells in blood
Arm/Group | Echinacea-based Dietary Supplement | Sugar Pill
Number analyzed (Participants) | 30 | 15
percent of red blood cells in blood | 41.5 (3.2) | 43.0 (3.6)

14. Secondary Outcome: Hematological Measures - Hematocrit
Description: as measured by hematocrit (Hct) at day 0 (baseline), day 14 (mid-intervention) and day 35 (post-intervention)
Time Frame: 35 days
Measure: Mean (Standard Deviation); unit: percent of red blood cells in blood
Arm/Group | Echinacea-based Dietary Supplement | Sugar Pill
Number analyzed (Participants) | 30 | 15
percent of red blood cells in blood | 44.5 (3.1) | 43.2 (3.6)

15. Secondary Outcome: Hematological Measures - Hemoglobin
Description: as measured by hemoglobin (Hb) at day 0 (baseline), day 14 (mid-intervention) and day 35 (post-intervention)
Time Frame: 0 days (baseline)
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Echinacea-based Dietary Supplement | Sugar Pill
Number analyzed (Participants) | 30 | 15
g/dL | 14.0 (1.2) | 14.7 (1.2)

16. Secondary Outcome: Hematological Measures - Hemoglobin
Description: as measured by hemoglobin (Hb) at day 0 (baseline), day 14 (mid-intervention) and day 35 (post-intervention)
Time Frame: 14 days (mid-intervention)
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Echinacea-based Dietary Supplement | Sugar Pill
Number analyzed (Participants) | 30 | 15
g/dL | 13.9 (1.1) | 14.6 (1.5)

17. Secondary Outcome: Hematological Measures - Hemoglobin
Description: as measured by hemoglobin (Hb) at day 0 (baseline), day 14 (mid-intervention) and day 35 (post-intervention)
Time Frame: 35 days
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Echinacea-based Dietary Supplement | Sugar Pill
Number analyzed (Participants) | 30 | 15
g/dL | 14.9 (1.2) | 14.5 (1.3)

ADVERSE EVENTS:
Time Frame: 35 days
Arm/Group | Echinacea-based Dietary Supplement | Sugar Pill
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/15
Other Adverse Events (participants affected / at risk) | 0/30 | 0/15

LIMITATIONS AND CAVEATS:
A limitation is that we did not control for the menstrual cycle. Additionally, we used self-reported physical activity data which relies on accuracy of reporting.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No